CLINICAL TRIAL: NCT06889402
Title: Risk Factors for Recurrence and Survival Outcomes of Esophageal Squamous Cell Carcinoma Patients with Complete Pathological Response After Neoadjuvant Therapy：A Multicenter Study
Brief Title: Prognostic Analysis of Esophageal Cancer with Complete Pathological Response After Neoadjuvant Therapy
Status: Not yet recruiting | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: AESCNT01
Record Dates: First submitted 2025-03-17; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2024-12

CONDITIONS: Esophageal Cancer
Keywords: Complete pathological response; neoadjuvant; Recurrence; Esophageal Squamous Cell Carcinoma; Survival
MeSH Terms: conditions — Esophageal Neoplasms; Pathologic Complete Response; Recurrence; Esophageal Squamous Cell Carcinoma | interventions — Neoadjuvant Therapy; Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- Recurrence: Patients with complete pathological response after neoadjuvant treatment experience recurrence or metastasis after surgery
  Interventions: Procedure: Neoadjuvant therapy with PD-L1 inhibitor
- Non-recurrence: Patients with complete pathological response after neoadjuvant treatment without recurrence or metastasis after surgery
  Interventions: Procedure: Neoadjuvant therapy with PD-L1 inhibitor

INTERVENTIONS:
Procedure: Neoadjuvant therapy with PD-L1 inhibitor — During neoadjuvant treatment, patients may receive neoadjuvant chemotherapy, neoadjuvant chemoradiotherapy, or neoadjuvant chemotherapy combined with immunotherapy during the perioperative period.
  Other Names: neoadjuvant chemotherapy; neoadjuvant chemoradiotherapy

SUMMARY:
Esophageal cancer is one of the most common malignant tumors worldwide, with high invasiveness and lethality. Currently, the treatment for resectable locally advanced esophageal cancer mainly consists of a treatment model centered on surgical treatment with the participation of multiple disciplines. Neoadjuvant treatment regimens include chemotherapy, chemoradiotherapy, and chemotherapy combined with immunotherapy. Complete pathological response (pCR)is currently regarded as one of the important indicators for evaluating the efficacy of neoadjuvant treatment. Previous studies have shown that 14%-39% of patients with complete pathological response after neoadjuvant treatment still experience recurrence and metastasis within two years after surgery, suggesting that pCR after esophageal cancer surgery does not mean clinical cure. Perhaps there is a highly risk clinical subgroup need to research. Therefore, based on the prospective clinical database of the National Cancer Center and in cooperation with multiple national cancer regional medical centers, this study analyzes and explores the prognosis of patients with locally advanced esophageal squamous cell carcinoma with pCR after neoadjuvant treatment, characterized by the Chinese population.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated neoadjvant treatment followed by esophagectomy from 2018 to 2023
* Patients with thoracic esophageal squamous cell carcinoma
* The preoperative clnical stage is cT1N+M0/cT2-4aN0-3M0, with potential resectability
* Patients with complete pathological response (ypT0N0M0)
* Without distant metastasis was found in the preoperative examinations, and the tumor did not directly invade the pancreas, spleen, trachea, aorta or other adjacent organs such as the lungs

Exclusion Criteria:

* Patients with previous history of malignant tumors
* Patients with multiple primary cancers
* Deficient neoadjuvant treatment or salvage surgery
* Incomplete clinical data

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with thoracic esophageal squamous cell carcinoma treated neoadjvant treatment followed by esophagectomy from 2018 to 2023,whose preoperative clnical stage was cT1N+M0/cT2-4aN0-3M0, with potential resectability and the ypstage ypT0N0M0（complete pathological response ）
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival | The postoperative follow-up period should last for at least one year.
  The time from the postoperative period of the patient to the first occurrence of recurrence or metastasis.

SECONDARY OUTCOMES:
Overall Survival Rate | The postoperative follow-up period should last for at least one year.
  the proportion of patients who are still alive for a certain period of time after surgery among all the patients who have undergone the surgical operation.

OTHER OUTCOMES:
Metastasis rate of different parts or organs | The postoperative follow-up period should last for at least one year.

CONTACTS AND LOCATIONS:
Locations (1):
- Section of Esophageal and Mediastinal Oncology, Department of Thoracic Surgery, National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No